CLINICAL TRIAL: NCT01825525
Title: Safety of the Colonoscope Magnetic Imaging Device (ScopeGuide®) in Patients With Implantable Cardiac Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Gareth Corbett, Specialist Registrar, Gastroenterology, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12/EE0075
Record Dates: First submitted 2013-04-03; First posted 2013-04-05 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cardiac device patients. (Experimental): Exposure to ScopeGuide - patients with cardiac devices exposed to ScopeGuide as per study protocol
  Interventions: Device: Exposure to ScopeGuide

INTERVENTIONS:
Device: Exposure to ScopeGuide — The 2 minute protocol exposure to the electromagnetic field of the ScopeGuide device.

SUMMARY:
The Olympus ScopeGuide® is a useful tool in speeding up colonoscopy and making it less painful for patients. It is currently contraindicated by the manufacturer for use with patients with implantable electronic devices (such as cardiac pacemakers). There is no evidence to back up this contraindication and with the number of pacemakers being inserted increasing by around 30 000 annually in the UK, more patients will be denied the use of this device should they require a colonoscopy.

Participants with Pacemakers or Implantable Cardioverter Defibrillators will attend their check appointment. Following this they will be asked to lie with a colonoscope connected to the ScopeGuide® placed onto their abdomen (with clothes on) for 2 minutes. During this time they will be monitored for any irregular cardiac activity which may indicate electromagnetic interference. After this a second device check will occur and the participant will be sent home.

The hypothesis is that the ScopeGuide will not interfere with the cardiac devices.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

Colonoscopy is the 'gold-standard' diagnostic procedure for visualising the inside of the large bowel. It involves the insertion of a flexible instrument called a "colonoscope" around the large bowel. During insertion, looping of the instrument inside the colon can lead to incomplete procedures and significant patient discomfort.

The development of the colonoscope magnetic imaging device (Olympus ScopeGuide®) has allowed the doctor performing the examination to detect looping of the instrument more easily. It has been shown in several studies that the duration, patient experience and completion rate of colonoscopy can be significantly improved by the use of ScopeGuide®.

The manufacturer advises against the use of ScopeGuide® for patients with implantable devices due to the theoretical hazard of electromagnetic interference leading to device malfunction. Therefore, patients with permanent pacemakers and implantable cardioverter-defibrillators (ICDs) who require colonoscopy are denied the potential benefits offered by ScopeGuide®. There is no documented evidence for this risk from case reports or studies and the investigators have used a simulator to demonstrate that ScopeGuide® caused no interference or malfunction.

The investigators propose an experimental study to evaluate the impact of the electromagnetic field created by ScopeGuide® on the implanted cardiac devices in patients. The study will be conducted in the Pacemaker Outpatient Clinic at Addenbrooke's hospital by a team of investigators including gastroenterologists and cardiologists. After giving their consent to participate, enrolled patients will have the activity of their cardiac device closely monitored while in close proximity to ScopeGuide® and any effect of this on the cardiac devices will be recorded.

The investigators hypothesise that ScopeGuide® does not create a magnetic field significant enough to interfere with the normal function of these devices. If true, patients with implanted cardiac devices can also be offered the benefit ScopeGuide® provides during colonoscopy.

The justification for this research is that the ScopeGuide® is currently not used in patients with implantable electronic cardiac devices (pacemakers and implantable cardioverter defibrillators(ICDs)) due to the manufacturers advice. There are no case reports and no studies in the medical literature to confirm or refute the advice and the investigators have demonstrated no evidence of interference using a simulator.

The number of patients with either a pacemaker or ICD is increasingly annually and with services such as the NHS bowel cancer screening programme in which colonoscopy is offered to patients with blood in their stool more of these patients are having this test.

To deny these patients the use of the ScopeGuide®, which has been shown to reduce procedure duration, reduce patient discomfort and increase completion rate without evidence is unjustified.

The investigators therefore believe that this project is justified to potentially allow patients with pacemakers or ICDs the benefit of ScopeGuide®. If the investigators demonstrate evidence of interference, it would demonstrate a lack of safety in this patient group.

Due to the lack of data for the safety of ScopeGuide® for patients with implantable cardiac devices we seek to question the current absolute contraindication imposed by the manufacturer. The main question to be answered by this study is whether implantable cardiac devices exhibit interference when exposed to the ScopeGuide®.

The population to be studied are individuals with implantable cardiac devices, attending their regular device check appointment at Addenbrooke's hospital. The age range will be 18 to 80 years. Those being studied will be able to give informed consent.

OBJECTIVES Primary Objective The primary objective of this study is to demonstrate in 100 serial participants whether the ScopeGuide® causes interference with implantable cardiac devices.

Secondary Objectives None STUDY DESIGN

Summary of Study Design

This study is an uncontrolled trial. The study method will be undertaken on 100 consecutive consenting participants.

The participants will be required for one visit only. This will be during their routine implantable device check appointment. Participation will extend their routine check appointment time by around 30 minutes. Once they have completed the study procedure they will not be required for follow up visits.

The duration of the study for an individual participant is as follows:

Attend regular cardiac device check appointment (around 20 minutes) Exposure to ScopeGuide® device while being monitored (around 10 minutes) Repeat cardiac device check (around 20 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Must have a permanent pacemaker or implantable cardioverter defibrillator
* Is attending for a routine pacemaker check during the study period

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Cardio-respiratory compromise on the day of the experiment (we propose NYHA Grade 3 or higher as criteria for this)
* Vulnerable adults

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Recruitment target met. | 6 to 8 months
  The study has a target recruitment of 100 patients. When this is met the study will stop.

SECONDARY OUTCOMES:
Interference seen with implanted cardiac device | 6 to 8 months
  If interference is seen in any of the recruited patients the study will be stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Ewen AB Cameron, MD MB ChB, Study Director — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Corbett GD, Lim YC, Lee JC, Chernolesskiy A, Pugh PJ, Cameron EA. Safety of the colonoscope magnetic imaging device (ScopeGuide) in patients with implantable cardiac devices. Endoscopy. 2014 Feb;46(2):135-8. doi: 10.1055/s-0033-1359044. Epub 2014 Jan 29. PMID 24477369